CLINICAL TRIAL: NCT04469439
Title: The Impact of Sinus Surgery in the Era of Highly Effective Modulatory Therapy
Brief Title: Impact of Sinus Surgery on Individuals With Cystic Fibrosis
Status: Recruiting | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Daniel M. Beswick, Assistant Professor-in-Residence, University of California, Los Angeles
Other Study IDs: 20-002079
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-07

CONDITIONS: Chronic Rhinosinusitis (Diagnosis); Cystic Fibrosis
Keywords: Chronic Rhinosinusitis; Cystic Fibrosis; Endoscopic Sinus Surgery
MeSH Terms: conditions — Disease; Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens are collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Surgical group: Individuals with cystic fibrosis and chronic rhinosinusitis who undergo endoscopic sinus surgery
- Medical group: Individuals with cystic fibrosis and chronic rhinosinusitis who do not undergo endoscopic sinus surgery

SUMMARY:
This study will be a prospective, observational study of patients who undergo endoscopic sinus surgery for cystic fibrosis-related chronic rhinosinusitis (CRS). Individuals who do not undergo surgery but are treated medically for CRS will also be enrolled to serve as a control group. Outcomes analyzed will include pulmonary, quality of life, and others.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects between the ages of 18 years old (inclusive) and 99 years old (inclusive, subjects over the age of 89 will be recorded to be 89 years old).
2. Diagnosed with cystic fibrosis as established by genetic testing combined with clinical assessment and/or sweat chloride
3. Diagnosed with chronic rhinosinusitis by multidisciplinary sinusitis guidelines
4. chronic rhinosinusitis symptoms persisting beyond initial medical treatment
5. Counseled for endoscopic sinus surgery and ongoing medical therapy with each patient electing their preferred treatment

Exclusion Criteria:

1. Underwent endoscopic sinus surgery in past 12 months
2. Will obtain follow up care at non-participating institutions
3. Unable to complete follow-up surveys

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from cystic fibrosis and otolaryngology outpatient clinics.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary function | baseline, 3, 6, 9, 12 months
  Pulmonary function will be measured using spirometry - the percent of predicted forced expiratory volume in the first second (ppFEV1)
Change in days of inpatient hospitalization | baseline, 3, 6, 9, 12 months
  Days of inpatient hospitalization will be assessed

SECONDARY OUTCOMES:
Change in quality of life | baseline, 3, 6, 9, 12 months
  Quality of life will be assessed using the 22-question SinoNasal Outcome test (range 0-110, with higher scores signifying worse quality of life)
Change in quality of life | baseline, 3, 6, 9, 12 months
  Quality of life will be assessed using the Cystic Fibrosis Questionnaire-Revised instrument (range 0-100, with higher scores signifying worse quality of life)
Change in olfaction | baseline, 3, 6, 9, 12 months
  Olfaction will be assessed using the Smell Identification Test (score range: 0-40, with higher scores demonstrated better olfactory ability)

OTHER OUTCOMES:
Patient satisfaction regarding treatment for chronic rhinosinusitis | at baseline
  Satisfaction will be assessed using 5-point Likert scales, ranging from 1 to 5 with 1 signifying "not important" and 5 signifying "very important"

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Beswick, MD, Principal Investigator — University of California, Los Angeles
Locations (9):
- United States (9):
  - University of California, Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - University of Colorado, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - University of North Carolina, Chapel Hill, North Carolina
  - Oregon Health Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Participant data will securely stored using REDCap software.

REFERENCES:
- [Derived] Liu CM, Fischer JL, Lee MJ, Mace JC, Kimple AJ, Markarian K, Alt JA, Bodner TE, Chowdhury NI, Chung SY, Eshaghian PH, Gao YA, Getz AE, Hwang PH, Khanwalkar A, Lee JT, Li DA, Norris M, Nayak JV, Overdevest JB, Owens C, Patel ZM, Pappas LE, Poch K, Schlosser RJ, Smith KA, Smith TL, Soler ZM, Suh JD, Turner GA, Wang MB, Taylor-Cousar JL, Saavedra MT, Beswick DM. Olfaction, Eating Preference, and Quality of Life in Cystic Fibrosis Chronic Rhinosinusitis. Laryngoscope. 2025 Jul;135(7):2476-2488. doi: 10.1002/lary.32155. Epub 2025 Mar 29. PMID 40156369
- [Derived] Liu CM, Fischer JL, Alt JA, Bodner TE, Chowdhury NI, Getz AE, Hwang PH, Kimple AJ, Mace JC, Smith TL, Soler ZM, Goss CH, Taylor-Cousar JL, Saavedra MT, Beswick DM. Impact of sinus surgery in people with cystic fibrosis and chronic rhinosinusitis in the era of highly effective modulator therapy: Protocol for a prospective observational study. PLoS One. 2024 Sep 26;19(9):e0310986. doi: 10.1371/journal.pone.0310986. eCollection 2024. PMID 39325787
- [Derived] Han EJ, Liu CM, Fischer JL, Mace JC, Markarian K, Alt JA, Bodner TE, Chowdhury NI, Eshaghian PH, Gao YA, Getz AE, Hwang PH, Khanwalkar A, Kimple AJ, Lee JT, Li DA, Norris M, Nayak JV, Owens C, Patel ZM, Poch K, Schlosser RJ, Smith KA, Smith TL, Soler ZM, Suh JD, Turner GA, Wang MB, Taylor-Cousar JL, Saavedra MT, Beswick DM. Impact of sociodemographic status and sex on chronic rhinosinusitis and olfaction in people with cystic fibrosis. Int Forum Allergy Rhinol. 2024 Nov;14(11):1700-1713. doi: 10.1002/alr.23402. Epub 2024 Jul 5. PMID 38967583